CLINICAL TRIAL: NCT03664986
Title: Pudendal Block Using Liposomal Bupivacaine vs. Standard Treatment During Sacrospinous Ligament Fixation: a Prospective Randomized Clinical Trial
Brief Title: Pudendal Block Using Liposomal Bupivacaine vs. Standard Treatment During Sacrospinous Ligament Fixation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Atlantic Health System (Other)
Responsible Party: Principal Investigator, Ricardo Caraballo, MD, Principal Investigator, Atlantic Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1191772
Record Dates: First submitted 2018-04-26; First posted 2018-09-11 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Vaginal Prolapse
MeSH Terms: conditions — Uterine Prolapse

STUDY DESIGN:
Who Masked: Participant
Masking Description: The group you get randomized to will be chosen by chance, like flipping a coin. Neither you nor the study doctor will choose what group you will be in. You will have an equal chance of being in either group. Neither you nor the nurses nor anesthesiologist will know which group you will be in. However, your study doctor will know.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exparel pudendal block (Experimental): This group will have intra-operative pudendal block performed with Liposomal Bupivacaine (EXPAREL) solution.
  Interventions: Drug: Liposomal Bupivacaine
- Comparison group (No Intervention): This group will be those to receive current standard treatment with no pudendal block performed.

INTERVENTIONS:
Drug: Liposomal Bupivacaine — The objective of our study is to compare the use of EXPAREL in minimizing post-operative pain after sacrospinous ligament fixation with or without concomitant procedures for pelvic organ prolapse, with or without suburethral sling. We hypothesize that pudendal nerve blockage using long-acting EXPAREL will reduce post-operative pain and potentially reduce oral narcotic consumption. It may also reduce the incidence of postoperative constipation and patient satisfaction.
  Other Names: Exparel
  Arms: Exparel pudendal block

SUMMARY:
A pudendal nerve block is a procedure where a local anesthetic is injected where the pudendal nerve is located. This allows quick pain relief to the perineum, vulva, and vagina. The purpose of this research study is see if injecting a long-acting local anesthetic, called Liposomal Bupivacaine (EXPAREL), will result in less post-operative pain after having vaginal prolapse surgery.

Typical post-operative pain lasts a few days. Short-acting anesthetics only provide pain relief in the few hours after surgery. EXPAREL will add the benefit of longer acting pain relief that can last up to 72 hours with the same safety profile. EXPAREL is an FDA-approved medication. It has been used and studied extensively in gynecologic surgery for incisional pain. It has also been studied in Urology and Orthopedic surgery with an excellent safety profile with good pain relief.

DETAILED DESCRIPTION:
Various clinical studies have indicated that preemptive analgesia can effectively reduce pain as well as analgesic requirements in the post-operative period. Pudendal nerve blockade has been used successfully for multiple urological procedures to prevent post-operative pain. It has also been used in obstetrical practice as a low-risk and low-cost anesthetic technique during repair of obstetrical lacerations.

Postoperative pain after vaginal reconstructive surgery is commonly localized to the vulva, lower vagina, and perineum, originating from the region of the sacrospinous ligament and pelvic floor. Therefore, pudendal nerve blockage has been employed safely during pelvic reconstructive surgery. A study comparing pudendal block with placebo after transvaginal reconstructive surgery did not produce any differences in post-operative pain intensity or the consumption of narcotic analgesia. However, the anesthetic used for the pudendal nerve blockage was short-acting non-liposomal bupivacaine with a half-life of 2.7 hours.

In 2011, a liposomal formulation of bupivacaine, EXPAREL, was approved by the FDA for single-dose infiltration in surgical site to produce postsurgical analgesia. The advantage of using this formulation of bupivacaine is that its analgesic effects can last up to 72 hours. Since the release of EXPAREL, there have been no published studies establishing its use for pudendal block or the management of postoperative pain in Urogynecologic surgery.

The objective of our study is to compare the use of EXPAREL in minimizing post-operative pain after sacrospinous ligament fixation with or without concomitant procedures for pelvic organ prolapse, with or without suburethral sling. We hypothesize that pudendal nerve blockage using long-acting EXPAREL will reduce post-operative pain and potentially reduce oral narcotic consumption. It may also reduce the incidence of postoperative constipation and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Female
* Able to give informed consent in English
* Electively scheduled for surgical management of pelvic organ prolapse involving sacrospinous ligament fixation

Exclusion Criteria:

* Pregnant or nursing
* Allergy to amide anesthetics
* History of opioid abuse
* Severe cardiovascular, hepatic, renal disease or neurological impairment
* Long-acting opioid within 30 days or any opioid use within 24 hours before surgery
* Patients taking monoamineoxidase inhibitors (MAOI) or antidepressants of the triptyline or imipramine types
* Administration of an investigational drug within 30 days before this study
* Chronic pain syndromes
* Daily NSAID or opioid use
* Contraindication to Non-steroidal anti-inflammatory drugs (NSAIDs)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2018-09-24 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain on postoperative day one | 24 hours post operative
  Pain on postoperative day one using the VAS (0 to 10 cm)

SECONDARY OUTCOMES:
Pain at the time of answering survey each day | Daily post-op days 1-3 and 7
  Pain at the time of answering survey each day [Time frame: post-operative days 1-3 and 7] using VAS (0 to 10 cm). (Self-reported via survey or telephone call)
Most intense pain each day | Daily post-op days 1-3 and 7
  Most intense pain each day [Time frame: post-operative days 1-3 and 7] using VAS (0 to 10 cm). (Self-reported via survey or telephone call)
Average pain each day | Daily post-op days 1-3 and 7
  Average pain each day [Time frame: post-operative days 1-3 and 7] using VAS (0 to 10 cm). (Self-reported via survey or telephone call)
Pain with sitting | Daily post-op days 1-3 and 7
  Pain with sitting [Time frame: post-operative days 1-3 and 7] using VAS (0 to 10 cm). (Self-reported via survey or telephone call)
Pain with first bowel movement | At time of first bowel movement
  Pain with first bowel movement using VAS (0 to 10 cm). (Self-reported via survey or telephone call)
Total narcotic consumption | up to 30 days post operative
  Total narcotic consumption
Urinary retention | up to 30 days post operative
  Incidence of Urinary Retention
Time to first bowel movement | up to 10 days post-operative
  Time to first bowel movement
Ambulatory Quality of Life questionnaire (QoR) | up to 24 hours before surgery and 72 hours post operative
  Quality of Life as measured by the ambulatory QoR [Time frame: pre-operative on the day of surgery and post-operative day 3].

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantic Health System, Morristown, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ezzedine D, Dhariwal L, Wasenda E, Salamon C, Caraballo R. Pudendal Nerve Block With Liposomal Bupivacaine for Sacrospinous Ligament Suspension. Urogynecology (Phila). 2024 Feb 1;30(2):98-106. doi: 10.1097/SPV.0000000000001397. Epub 2023 Jul 13. PMID 37450670